CLINICAL TRIAL: NCT02552264
Title: Implementing and Evaluating an Empirically Supported Training Program to Enhance Emotional Management Skills and Professional Resiliency in Healthcare Providers
Brief Title: Testing a Training Program to Enhance Emotional Management Skills and Professional Resiliency in Healthcare Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: IWK Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NSHA REB ROMEO File #: 1019748
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Burnout, Professional; Adaptation, Psychological
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention (Active Comparator): Acceptance and Commitment Therapy
  Interventions: Behavioral: Acceptance and Commitment Therapy for the Workplace
- Waitlist control (Placebo Comparator): Acceptance and Commitment Therapy
  Interventions: Behavioral: Acceptance and Commitment Therapy for the Workplace

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy for the Workplace — Acceptance and Commitment Therapy
  Other Names: Professional Resiliency

SUMMARY:
The Behaviour Change Institute (BCI) was created in 2008 within Capital Health to provide healthcare providers with evidence-based skills in helping patients change. In addition, the BCI has also become a resource within the organization to assist with other needed changes, such as helping healthcare providers use new or different procedures to provide better patient care. Through our work at the BCI we have identified the need to help healthcare providers to better cope with change. The purpose of this project is to implement and to evaluate an evidence-based professional resiliency training program for staff to help them better cope with change. This professional resiliency training program is based on an empirically supported form of therapy called Acceptance and Commitment Therapy. The training takes the form of a hands-on, applied workshop designed to increase resiliency and flexibility in a workplace setting.

DETAILED DESCRIPTION:
The Behaviour Change Institute (BCI) was created in 2008 within Capital Health to provide healthcare providers with behaviour change counselling skills. These skills are backed by evidence-based theory and competency training methods and are designed to be used by healthcare providers to help their patients change their behaviours. Acquiring these skills involves change for the healthcare provider. Through our work at the BCI we have come to identify the need to help healthcare providers effectively manage their emotions in such situations in order to learn behavior change counselling skills and to continue to use them effectively over time. The ability to effectively manage emotions, including discomfort and distress, may differentiate between individuals who are able to successfully adopt and maintain new behaviours over time from those who do not (Brown, Lejuez, Kahler, Strong, & Zvolensky, 2005). That is, we have identified that there is a significant need to support healthcare providers to more effectively manage emotions in order to help them change.

The Acceptance and Commitment Therapy for the Workplace program (ACT-W) is an evidence-based program designed to help individuals manage emotions and stress by learning skills to accept negative feelings, thoughts, and sensations and to move toward valued behaviours (Flaxman, Bond, Livheim, Hayes, 2013). The ACT-W program has been shown to increase the ability to manage emotions and stress (Flaxman & Bond, 2010) and to increase the ability to learn new behaviours (Bond & Flaxman, 2006; Luoma et al., 2007; Varra, Hayes et al., 2008).

The purpose of this project is to evaluate the implementation of the ACT-W training program for healthcare providers through the BCI.

ELIGIBILITY:
Inclusion Criteria:

* Employees (full time or part time; administrative or clinical) within service areas with managerial approval to attend the training program.

Exclusion Criteria:

* None

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Psychological Flexibility | Change from T1 (baseline) to T2 (1 week) and change from T1 (baseline) to T3 (3 months)
  The Acceptance and Action Questionnaire, a 7-item self-report scale which measures one's willingness to experience difficult thoughts and emotions while also persisting in the pursuit of values and goals.

SECONDARY OUTCOMES:
Change in Burnout | Change from T1 (baseline) to T2 (1 week) and change from T1 (baseline) to T3 (3 months)
  The Maslach Burnout Inventory, a 22-item self-report scale that measures three facets of burnout including emotional exhaustion (e.g. emotionally overextended within one's job); depersonalization (e.g. having impersonal responses to one's customers/clients; and personal accomplishment (e.g. sense of competence).
Absenteeism | at 2 years
  Number of hours missed from the workplace due to illness from time sheets submitted by each employee to payroll.

CONTACTS AND LOCATIONS:
Overall Officials: Dayna Lee-Baggley, Ph.D., Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada